CLINICAL TRIAL: NCT03290794
Title: Structured Post-marketing Surveillance to Collect the Safety Data of Intravitreal Aflibercept Injection (IVT-AFL) in Patients of Wet Age-related Macular Degeneration During Real World Clinical Practice
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19140
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Wet Age-related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Decision to treat with intravitreal aflibercept for wet AMD: Adult patients with a diagnosis of wet AMD, as an indication approved by the local health authorities for use with intravitreal aflibercept.
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, BAY86-5321) — Intravitreal Aflibercept as prescribed by the treating Physician

SUMMARY:
The proposed regulatory post-marketing surveillance (PMS) study will be planned to collect the safety data of aflibercept intravitreal injection in patients with wet Age-related Macular Degeneration (AMD) in real-life treatment practice

The primary objective is:

- To collect safety data in wet AMD patients treated with intravitreal aflibercept injection

The secondary objective is:

- To determine how disease activity is monitored including type and frequency of ocular tests and frequency of injections

DETAILED DESCRIPTION:
The study will be multicenter, observational, prospective, single arm, post marketing surveillance study of intravitreal aflibercept injection in wet AMD patients in routine clinical practice and real-life conditions without any protocol mandated interventions.

Approximately 100 wet AMD patients from up to ten ophthalmology clinics across India will be enrolled in this study. Each study site will be requested to enroll approximately 10 patients, however, the sites will be asked to enrolled additional patients in case of failure to enroll 10 patients by other site to complete the recruitment of approximately 100 patients.

Patients will be observed for maximum period of 6 months after the start of intravitreal aflibercept treatment. The observation period should cover the entire period from initial visit to the last follow-up visit at six months or withdrawal of consent, or the patient is lost to follow up (whatever is earliest).

The study site will be asked to enroll into the study all consecutive patients with wet AMD for whom the decision has been made to treat with intravitreal aflibercept injection and patients agrees to sign informed consent form for data collection purpose.

Any switch to another therapy or initiated administration of other anti-VEGF (Vascular Endothelial Growth Factor) injection in fellow eye or the discontinuation of treatment with IVT-AFL before the 6 month implies the end of the observation period. However, the safety follow-up will continue at least 30 days after last intravitreal aflibercept injection or in case of the discontinuation of treatment with IVT-AFL or till the patient switch the treatment from IVT-AFL and received other anti-VEGF injection before the 6 month observation period.

ELIGIBILITY:
Inclusion Criteria:

* Decision to treat with intravitreal aflibercept injection prior to patient enrolment as per the treating ophthalmologist's routine clinical practice.
* Adult patients with a diagnosis of wet AMD, as an indication approved by the local health authorities (DCGI) for use with intravitreal aflibercept injection.
* Patient or legal delegate signed informed consent.

Exclusion Criteria:

* Participation in a clinical trial of an investigational agent within 30 days.
* Patients receiving other anti-VEGF agent in fellow eye.
* Contraindications according to the local prescribing information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously treated with any systemic or other intravitreal anti-VEGF treatment will be included in this study after the window period of 30 days to avoid the risks of unknown additive effects that might be associated with previous anti-VEGF treatments .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Frequency of reported ocular and non-ocular adverse events during observation period | Up to 6 months
  unilateral / bilateral treatment
Percentage of reported ocular and non-ocular adverse events during observation period | Up to 6 months
  unilateral / bilateral treatment

SECONDARY OUTCOMES:
Type of ocular tests undertaken | Up to 6 months
  e.g. Visual acuity, ocular computed tomography, indocyanine angiography, Angiography, Fundus photography
Interval between ocular test | Up to 6 months
  Date of ocular test
Date of aflibercept injections | Up to 6 months
  Date of aflibercept injections
Injection dose | Up to 6 months
  Injection dose
Interval (days) between aflibercept injections | Up to 6 months
  During observation periods
Frequency of monitoring / clinic visits | Up to 6 months
  Frequency of monitoring / clinic visits

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, India

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/